CLINICAL TRIAL: NCT06567236
Title: E4D Compare Adapted to Evaluate Pulpal Access Cavity Preparation in the D2 Preclinical Endodontics Course: Educational Randomized Controlled Trial
Brief Title: E4D Compare Adapted to Preclinical Endodontics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB2022-1492-CD-EXM
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Self-Assessment; Self-Perception
Keywords: Endodontics; Predental education; Educational technology; Teaching methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional teaching method (No Intervention): Participants will be exposed to traditional teaching method.
- 3D software teaching method. (Experimental): Participants will be exposed to traditional teaching method and 3D software teaching method.
  Interventions: Other: 3D software

INTERVENTIONS:
Other: 3D software — Participants in the experimental arm will receive extra training on Planmeca Romexis Compare Software adapted to evaluate endodontic access preparation.
  Arms: 3D software teaching method.

SUMMARY:
Based on pilot study's promising results, we decided to further investigate the impact of adapting Planmeca Romexis Compare software to evaluate pulpal access preparations on second-year dental students' technical performance, self-evaluation skills and opinions. No educational records, grades, coursework, or any other assignments that are completed as part of the regular class will be analyzed as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Second-year dental students enrolled in DDDS 719 Integrated Practice of Dentistry Lab II during 2022-2023 at Texas A&M School of Dentistry
* Students who have completed fixed prosthodontics preclinical course
* Students attending the endodontics preclinical course.

Exclusion Criteria:

* First, third and fourth-year dental students at Texas A&M School of Dentistry
* Second-year dental students NOT enrolled in DDDS 719 Integrated Practice of Dentistry Lab II during 2022-2023 at Texas A&M School of Dentistry
* Students who are not interested in participating.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Self-assessment - traditional method vs traditional method plus 3D software method | baseline, 2 weeks, 4 weeks, 5 weeks and 7 weeks
  Compare self-assessment after traditional method only and with extra 3D software method
Grading - traditional method vs traditional method plus 3D software method | baseline, 2 weeks, 4 weeks, 5 weeks and 7 weeks
  Compare technical skills after traditional method only and with extra 3D software method

SECONDARY OUTCOMES:
Grading - traditional/visual grading vs 3D software grading | baseline, 2 weeks, 4 weeks, 5 weeks and 7 weeks
  Compare traditional/visual grading to 3D software grading using different tolerance levels

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M School of Dentistry, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poly A, Burnett JE, Buie CA, Schweitzer JL. Three-dimensional software adapted to evaluate endodontic access cavity preparation. J Dent Educ. 2023 Dec;87 Suppl 3:1848-1851. doi: 10.1002/jdd.13216. Epub 2023 Apr 11. No abstract available. PMID 37016471